CLINICAL TRIAL: NCT00897312
Title: Title: Evaluation of Systemic IDO Levels After Various Immunotherapeutics
Brief Title: Effect of Biological Therapy on Biomarkers in Patients With Untreated Hepatitis C, Metastatic Melanoma, or Crohn Disease
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey A. Sosman, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC MEL0651; VU-VICC-MEL-0651; VU-VICC-060614
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma
Keywords: stage IV melanoma; hepatitis C infection; melanoma (skin); precancerous/nonmalignant condition
MeSH Terms: conditions — Melanoma; Hepatitis C; Precancerous Conditions | interventions — Infliximab; tremelimumab; Ribavirin; Chromatography, High Pressure Liquid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Serum/plasma samples will be collected from patients being treated for untreated acute and chronic Hepatitis C with pegylated IFN-α and ribavirin
  * Serum/plasma samples will be collected from patients being treated for metastatic melanoma with CYP-206,675
  * Serum/plasma samples previously collected
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: infliximab
  Other Names: Remicade
Biological: pegylated interferon alfa
  Other Names: pegylated interferon-a
Biological: ticilimumab
  Other Names: CP-675206
Drug: ribavirin
  Other Names: Copegus, Rebetol, Ribasphere
Other: high performance liquid chromatography
  Other Names: not noted
Other: laboratory biomarker analysis
  Other Names: not noted

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer, hepatitis C, or Crohn disease in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer and other diseases.

PURPOSE: This laboratory study is looking at the effect of biological therapy on biomarkers in patients with untreated hepatitis C, metastatic melanoma, or Crohn disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine how a variety of immune-modulating therapies (i.e., interferon alfa [IFN-α] in patients with untreated acute or chronic hepatitis C, anti-tumor necrosis factor in patients with active inflammatory bowel disease (i.e., Crohn disease), and anticytotoxic T-lymphocyte antigen immunoglobulin in patients with metastatic melanoma) affect the tissue expression of indoleamine 2, 3 dioxygenase (IDO), a major immune-regulatory mechanism.
* To determine whether administration of pegylated INF-α in patients with untreated acute and chronic hepatitis C causes systemic changes in the IDO pathway, as indicated by lowered serum tryptophan (TRP) and elevated serum kynurenine (KYN).
* To determine whether administration of ticilimumab (i.e., anti-CTLA4 human monoclonal antibody CP-675,206) in patients with metastatic melanoma inhibits activation of the IDO pathway as indicated by normal serum TRP and normal serum KYN.
* To determine whether administration of infliximab in patients with Crohn disease inhibits activation of the IDO pathway, as indicated by normal serum TRP and normal serum KYN.

OUTLINE: Serum samples are collected from patients with hepatitis C and metastatic melanoma at baseline and at 3 to 4 weeks after treatment is initiated. Previously collected samples from patients with Crohn disease are also assessed at these time points. Samples are analyzed for tryptophan and kynurenine levels via high-performance liquid chromatography.

PROJECTED ACCRUAL: A total of 15 patients with untreated acute or chronic Hepatitis C, 15 patients with metastatic melanoma, and 20 patients with Crohn disease will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute or chronic hepatitis C

    * Receiving pegylated interferon alfa and ribavirin
  * Metastatic melanoma

    * Receiving ticilimumab
  * Crohn disease

    * Received prior infliximab

Exclusion Criteria:

* Not specified

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with Hepatitis C; Anti-TNF in patients with active inflammatory bowel disease(IBD); anti-CTLA Ig in patients with metastatic melanoma
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Systemic indoleamine 2, 3 dioxygenase levels in tissue at baseline and 3 to 4 weeks after treatment is initiated (timepoints for cancer and hepatitis patients) | at baseline and 3 to 4 weeks after treatment is initiated
Serum TRP levels at baseline and at 3 to 4 weeks after treatment is initiated (timepoints for cancer and hepatitis patients) | at baseline and at 3 to 4 weeks after treatment is initiated
Serum KYN levels at baseline and at 3 to 4 weeks after treatment is initiated (timepoints for cancer and hepatitis patients) | at baseline and at 3 to 4 weeks after treatment is initiated

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Sosman, MD, Study Chair — Vanderbilt-Ingram Cancer Center